CLINICAL TRIAL: NCT00955890
Title: Randomized Phase II Trial Of Interventional Therapy Investigate Cardiac Protection of Dexrazoxane In Women With Breast Cancer Having Experienced Grade 1 Cardiotoxicity During Prior Anthracycline-based Chemotherapy.
Brief Title: Dexrazoxane as a Protective Agent in Anthracycline Treated Breast Cancer
Acronym: cardioprotec
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrolled too slow
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xichun Hu, Dr, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MBC0901 FUCH
Record Dates: First submitted 2009-08-07; First posted 2009-08-10 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Breast Cancer
Keywords: cardioprotection; anthracycline chemotherapy; breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Dexrazoxane; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- control arm (No Intervention): anthracycline chemotherapy only
- low dose dexrazoxane group (Experimental): anthracycline chemotherapy plus low dose dexrazoxane(10:1)
  Interventions: Drug: Dexrazoxane hydrochloride
- middle dose dexrazoxane group (Experimental): anthracycline chemotherapy plus middle dose dexrazoxane(15:1)
  Interventions: Drug: Dexrazoxane hydrochloride

INTERVENTIONS:
Drug: Dexrazoxane hydrochloride — pink power 250mg/bottle DEX:EPI,10:1 every 3 weeks
  Other Names: Dexrazoxane for Injection
  Arms: low dose dexrazoxane group; middle dose dexrazoxane group
Drug: Dexrazoxane hydrochloride — pink powder 250mg/bottle DEX:EPI,15:1 every 3 weeks
  Other Names: dexrazoxane injection
  Arms: middle dose dexrazoxane group

SUMMARY:
Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Chemoprotective drugs, such as dexrazoxane, may protect normal cells from the side effects of chemotherapy. Monoclonal antibodies such as trastuzumab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Radiation therapy uses high-energy x-rays to damage tumor cells. CTnT/cTnI/ANP/BNP were proved to be used as a biomarker of drug related cardiotoxicity. There are excellent correlations between the total cumulative dose of doxorubicin, the severity of the resulting cardiomyopathy, and the level of serum troponin-T.

DETAILED DESCRIPTION:
Patients with breast cancer receiving anthracycline chemotherapy randomized to 3 groups:chemotherapy plus low dose dexrazoxane,chemotherapy plus middle dose dexrazoxane, chemotherapy only.Every patient receive at least 2 cycles anthracycline chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

DISEASE CHARACTERISTICS:

* Histologically confirmed primary infiltrating adenocarcinoma of the breast

  * Confirmed by core needle biopsy or incisional biopsy or surgery
  * Experienced grade 1 cardiac toxicity during prior anthracycline-based chemotherapy
  * At least 2 cycles same anthracycline based chemotherapy are needed

Exclusion Criteria:

* Accumulated dose of EPI ≥1000mg/m2,ADM≥550mg/m2
* With the following risk factors: Uncontrolled or severe cardiovascular disease (e.g., myocardial infarction within the past 6 months, congestive heart failure treated with medications, or uncontrolled hypertension); Prior or Concurrent radiation to heart
* Pregnant or nursing
* Other currently active malignancy except nonmelanoma skin cancer
* Uncontrolled or severe bleeding,diarrhea,intestinal obstruction
* Grade 2 or more Cardiac Toxicity (CTC AE3.0)

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-06; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Occurence of cardiac toxicity in patients with breast cancer receiving anthracycline chemotherapy | 1 year

SECONDARY OUTCOMES:
Relationship between serum level of cTnT/cTnI/ANP/BNP and cardiac toxicity | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: xichun Hu, MD, Principal Investigator — member of Fudan University
Locations (1):
- Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China